CLINICAL TRIAL: NCT04303689
Title: Repurposing Colchicine to Improve Vascular Function in Hypertension
Acronym: RECTIFHY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: University of Aarhus (Other)
Responsible Party: Principal Investigator, Ylva Hellsten, Professor, Dr. Med. Sc., University of Copenhagen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: Colchicine study
Record Dates: First submitted 2020-01-23; First posted 2020-03-11 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Essential Hypertension
Keywords: essential hypertension; colchicine; vascular function; vascular compliance; blood pressure
MeSH Terms: conditions — Essential Hypertension | interventions — Colchicine

STUDY DESIGN:
Intervention Model Description: Single blinded randomized placebo-controlled intervention
Who Masked: Participant
Masking Description: Subjects are blinded and randomized to receive either colchicine-treatment or placebo
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Colchicine (Experimental): 3 weeks of treatment with colchicine
  Interventions: Drug: Colchicine Tablets
- Placebo (Placebo Comparator): 3 weeks of placebo-treatment
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Colchicine Tablets — patients with essential hypertension are randomized to receive either 3 weeks of colchicine
  Other Names: Colchicine
  Arms: Colchicine
Drug: Placebo — patients with essential hypertension are randomized to receive either 3 weeks of placebo-treatment
  Arms: Placebo

SUMMARY:
In this project the potential beneficial effect of the drug colchicine on vascular reactivity and blood pressure will be assessed. Colchicine is a commonly used anti-inflammatory medication approved for the treatment of gout, Familial Mediterranean Fever and pericarditis in Denmark. The current project idea is based on accumulating evidence in the literature for a beneficial role of colchicine treatment in the prevention of cardiovascular disease in parallel with novel mechanistic insight from our own research. Recently, colchicine was associated with a lower risk of cardiovascular disease, including reduced myocardial infarctions, strokes and acute coronary syndrome . However, none of these trials have investigated the effect of colchicine on arterial tone or stiffness, changes to which may underlie the reduced risk of cardiovascular disease associated with colchicine. In support of the hypothesis that colchicine will improve vascular reactivity, a study in 1985 by Lagrue et al. found that daily, low-dose colchicine improved arterial stiffness in a small cohort of hypertensive patients. More recently, colchicine was shown to improve arterial stiffness in patients with Familial Mediterranean fever supporting a cardiovascular protective role of colchicine. Finally, colchicine is also proposed to have anti-inflammatory effects in the vascular system.

DETAILED DESCRIPTION:
In this project w the potential beneficial effect of the drug colchicine on vascular reactivity and blood pressure is evaluated. Colchicine is a commonly used anti-inflammatory medication approved for the treatment of gout, Familial Mediterranean Fever and pericarditis in Denmark. The current project idea is based on accumulating evidence in the literature for a beneficial role of colchicine treatment in the prevention of cardiovascular disease in parallel with novel mechanistic insight from research of the investigators. Recently, colchicine was associated with a lower risk of cardiovascular disease, including reduced myocardial infarctions, strokes and acute coronary syndrome. However, none of these trials have investigated the effect of colchicine on arterial tone or stiffness, changes to which may underlie the reduced risk of cardiovascular disease associated with colchicine. In support of thehypothesis that colchicine will improve vascular reactivity, a study in 1985 by Lagrue et al. found that daily, low-dose colchicine improved arterial stiffness in a small cohort of hypertensive patients. More recently, colchicine was shown to improve arterial stiffness in patients with Familial Mediterranean fever supporting a cardiovascular protective role of colchicine. Finally, colchicine is also proposed to have anti-inflammatory effects in the vascular system.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with essential hypertension
* BMI<30
* blood pressure (sys/dia) ≥120 mmhg and/or ≥80 mmhg while on hypertensive medication OR
* blood pressure (sys/dia) ≥130 mmhg and/or ≥85 mmhg without hypertensive medication

Exclusion Criteria:

* smoking
* excessive alcohol use
* chronic diseases (beside essential hypertension)

Ages: 40 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Changes in vascular function with treatment measured as flowchanges with ultrasound doppler in response to infusions of isoprenaline | Change in vascular conductance in response to infusions is assessed after acute treatment and before and within 72 hours after the 3 weeks of colchicine or placebo treatment
  Infusions of isoprenalin in the brachial artery, measurement of blood flow with ultrasound doppler and intraarterial blood pressure with an intraarterial transducer for the calculation of leg vascular conductance
Changes in vascular function with training measured as flowchanges with ultrasound doppler divided by changes in blood pressure measured with intraarterial canula, in response to infusions of acetylcholine | Change in vascular conductance in response to infusions is assessed after acute treatment before and within 72 hours after the 3 weeks of colchicine or placebo treatment
  Infusions of acetylcholine in the brachial artery, measurement of blood flow with ultrasound doppler and intraarterial blood pressure with an intraarterial transducer for the calculation of leg vascular conductance
Changes in vascular function with training measured as flowchanges with ultrasound doppler divided by changes in blood pressure measured with intraarterial canula, in response to infusions of sodium nitroprusside | Change in vascular conductance in response to infusions is assessed after acute treatment and before and within 72 hours after the 3 weeks of colchicine or placebo treatment
  Infusions of sodium nitroprusside in the brachial artery, measurement of blood flow with ultrasound doppler and intraarterial blood pressure with an intraarterial transducer for the calculation of leg vascular conductance

SECONDARY OUTCOMES:
Blood pressure | Measurements are made before and after 3 weeks of treatment with colchicine or placebo.
  Blood pressure measured at home with an automated blood pressure device
Vascular compliance | Measurements are made before and after 3 weeks of treatment with colchicine or placebo.
  measured by intraarterial blood pressure and changes in arterial diameter by ultrasound doppler

CONTACTS AND LOCATIONS:
Overall Officials: Ylva Hellsten, Dr. Med. Sc., Principal Investigator — University of Copenhagen
Locations (1):
- Department of Nutrition, Exercise and Sports, UCopenhagen, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ehlers TS, van der Horst J, Moller S, Piil PK, Gliemann L, Aalkjaer C, Jepps TA, Hellsten Y. Colchicine enhances beta adrenoceptor-mediated vasodilation in men with essential hypertension. Br J Clin Pharmacol. 2023 Jul;89(7):2179-2189. doi: 10.1111/bcp.15688. Epub 2023 Feb 24. PMID 36764326